CLINICAL TRIAL: NCT04879095
Title: Urdu Translation, Validity and Reliability of Dyspnea 12 (D-12)
Status: Completed | Type: Observational
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Other Study IDs: REC00780 Mehwish Shabbir
Record Dates: First submitted 2021-05-04; First posted 2021-05-10 (Actual); Last update posted 2021-06-29 (Actual); Status verified 2021-06

CONDITIONS: COPD
Keywords: Body mass index (BMI); Rate of perceived exertion (RPE); 6 minute walk test (^MWT)
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Dyspnea is a distressing symptom with pain like perception. The object of study is to translate a tool that measure overall dyspnea severity. Although many scales are available to assess dyspnea but D12 is a clear reliable scale and is use full in clinical practice to assess dyspnea in terms of intensity, quality and emotional response.

DETAILED DESCRIPTION:
Aim of study is to translate a clinical validate of Urdu version of D-12 in COPDs patients. The study will measure reliability & validity of dyspnea in Urdu version. No study has been conducted in our region to translate D-12 follow the proper cross culture adaptation. Therefor the instrument will translate in our language adapting proper cross culture guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Patient age between 40-65 with diagnosis of COPD
* Outpatient individual who are on follow up
* Healthy individual
* Those who can read and understand English and Urdu as well.

Exclusion Criteria:

* Patient with cognitive impairment or sensory disorder were exclude.
* Patient physical disability
* Refuse to perform test

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: COPD
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2020-08-13 (Actual); Primary Completion 2021-04-24 (Actual); Study Completion 2021-04-24 (Actual)

PRIMARY OUTCOMES:
Translation of Dyspnea 12 in Urdu version | 4 Week
  D12 scale is used in assessment of dyspnea severity using its descriptors consist of sensory quality and effective component. It's a 12 item scale from 1-7 item related to physical component score (quality of sensation of dyspnea) & from 8-12 related to emotional response of this sensation. Each item was graded on 4 point scale as none, mild, moderate & severe and scored as 0 to 3 to get final score of 0 to 36
  * Forward conversion
  * Professional panel
  * Backward conversion
  * Pretesting
  * Final Form The translation of Dyspnea12 (D-12) Questionnaire into Urdu was done by using Cross Cultural Adaptation techniques according to WHO guideline it involve the following steps
  * Forward conversion
  * Professional panel
  * Backward conversion
  * Pretesting
  * Final Form

SECONDARY OUTCOMES:
Six minute Walk test | 4 week
  It is a sub-maximal exercise test used to assess aerobic capacity and endurance. The distance covered over a time of 6 minutes is used as outcome by which to compare changes in performance capacity. 30-metre stretch of unimpeded walkway is used and patient is instructed to walk as far as possible for 6 minutes. Test retest reliability of 6MWT showed good internal consistency (ICC=0.9) in patients with heart failure patients
Rate Perceived Exertion | 4 week
  The scale is used to monitor and guide exercise intensity and help in measure how hard your body is working when you exercise. It gives estimate of your heart rate and exercise intensity zone. The scale ranges from 6 -20. 6 indicate no exertion and 20 denotes maximum exertion, it is simple numerical list.

CONTACTS AND LOCATIONS:
Overall Officials: sumaiyah Obaid, MS, Principal Investigator — Riphah International University
Locations (1):
- Civil Hospital, Hyderābād, Sindh, Pakistan